CLINICAL TRIAL: NCT01041170
Title: Antagonist-Elicited Cannabis Withdrawal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 999906410; 06-DA-N410
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-01-11

CONDITIONS: Cannabis; Dependence
Keywords: Rimonabant; fMRI; Alternative Matrices; Brain Imaging; THC
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; Rimonabant

INTERVENTIONS:
Drug: THC
Drug: Rimonobant
Drug: Rimonabant

SUMMARY:
Background: Rimonabant, a CB1 receptor antagonist, blocks effects of cannabinoids and, in dependent animals, elicits cannabinoid withdrawal. No studies have examined rimonabantelicited cannabis withdrawal in humans.

Goals: (1) Determine the lowest single dose of oral rimonabant that elicits measurable cannabinoid withdrawal. (2) Characterize cognitive performance, subjective state, physiological condition, and regional brain activation (measured by functional magnetic resonance imaging [fMRI]) during acute and chronic administration of oral delta 9-tetrahydrocannabinol (THC) and during cannabis withdrawal. (3) Characterize the pharmacokinetics of oral THC and metabolites in body fluids and hair and of rimonabant in plasma.

Subject Population: Up to 60 completing cannabis users aged 18-45 (up to 24 in Experiment I, 36 in Experiment II) and 18 completing non-drug-using controls (Experiment II). Enrollment target is 82% Caucasian, 14% African American, 4% other; 9% Hispanic; 35% women.

Experimental Design and Methods: Experiment I: In this within-subject, randomized, double-blind, dose-escalation study, six participants receive 7 days of THC (40-120 mg/day). On Day 8, five participants receive 20 mg rimonabant; one receives placebo. If withdrawal criteria (greater than or equal to 150% or 2.5-fold increase in selected visual-analog scales) are not met in all five participants receiving rimonabant, separate groups of six are similarly treated with 40, 60 or 80 mg rimonabant, if necessary. The PI and MRP will submit all adverse events and relevant cardiovascular and scientific data to the IRB at the completion of each rimonabant dose panel. When the extramural NIDA DSMB is in place, it will review all data collected to date and develop and implement a monitoring plan, including review on completion of each dose cohort. DSMB recommendations will be reviewed by the Sponsor, Clinical Director and IRB before proceeding to the next dose cohort. In addition, if any subject has an intolerable adverse event (ie, an adverse event leading to study discontinuation) or serious adverse event in response to rimonabant on Day 8, the blind for that subject will be broken, and a report sent to the Sponsor, the extramural NIDA DSMB when in place and the IRB for discussion.

Experiment II: In this randomized, placebo-controlled, double-blind study, 36 participants receive 7 days of THC (40-120 mg/day). On Day 8, 18 participants receive rimonabant dose determined in Experiment I to elicit cannabis withdrawal; 18 participants receive placebo rimonabant to evaluate spontaneous cannabis withdrawal. Cognitive, psychological, physiological and hormonal measures are monitored to determine onset, magnitude, and duration of THC intoxication and withdrawal and to correlate with THC and rimonabant pharmacokinetics. Changes in blood oxygen level-dependent (BOLD) signal are determined with five fMRI scans throughout the study. Eighteen non-drug-using controls undergo scanning and cognitive testing at similar intervals.

Risks and Benefits: The proposed doses of THC and rimonabant have been well tolerated in other studies. The most common side effects of oral THC are sedation, cognitive impairment, euphoria, poor coordination, tachycardia, and hypotension. Spontaneous withdrawal from cannabis is mild and medically benign. Experience with other drugs suggests that antagonist-elicited cannabis withdrawal may have an earlier onset and greater intensity than spontaneous cannabis withdrawal. There are no clinical benefits to participants. Scientific benefits are greater understanding of cannabis intoxication, tolerance, and withdrawal and of the role of rimonabant in eliciting cannabis withdrawal.

DETAILED DESCRIPTION:
Background: Rimonabant, a CB1 receptor antagonist, blocks effects of cannabinoids and, in dependent animals, elicits cannabinoid withdrawal. No studies have examined rimonabantelicited cannabis withdrawal in humans.

Goals: (1) Determine the lowest single dose of oral rimonabant that elicits measurable cannabinoid withdrawal. (2) Characterize cognitive performance, subjective state, physiological condition, and regional brain activation (measured by functional magnetic resonance imaging [fMRI]) during acute and chronic administration of oral delta 9-tetrahydrocannabinol (THC) and during cannabis withdrawal. (3) Characterize the pharmacokinetics of oral THC and metabolites in body fluids and hair and of rimonabant in plasma.

Subject Population: Up to 60 completing cannabis users aged 18-45 (up to 24 in Experiment I, 36 in Experiment II) and 18 completing non-drug-using controls (Experiment II). Enrollment target is 82% Caucasian, 14% African American, 4% other; 9% Hispanic; 35% women.

Experimental Design and Methods: Experiment I: In this within-subject, randomized, double-blind, dose-escalation study, six participants receive 7 days of THC (40-120 mg/day). On Day 8, five participants receive 20 mg rimonabant; one receives placebo. If withdrawal criteria (greater than or equal to 150% or 2.5-fold increase in selected visual-analog scales) are not met in all five participants receiving rimonabant, separate groups of six are similarly treated with 40, 60 or 80 mg rimonabant, if necessary. The PI and MRP will submit all adverse events and relevant cardiovascular and scientific data to the IRB at the completion of each rimonabant dose panel. When the extramural NIDA DSMB is in place, it will review all data collected to date and develop and implement a monitoring plan, including review on completion of each dose cohort. DSMB recommendations will be reviewed by the Sponsor, Clinical Director and IRB before proceeding to the next dose cohort. In addition, if any subject has an intolerable adverse event (ie, an adverse event leading to study discontinuation) or serious adverse event in response to rimonabant on Day 8, the blind for that subject will be broken, and a report sent to the Sponsor, the extramural NIDA DSMB when in place and the IRB for discussion.

Experiment II: In this randomized, placebo-controlled, double-blind study, 36 participants receive 7 days of THC (40-120 mg/day). On Day 8, 18 participants receive rimonabant dose determined in Experiment I to elicit cannabis withdrawal; 18 participants receive placebo rimonabant to evaluate spontaneous cannabis withdrawal. Cognitive, psychological, physiological and hormonal measures are monitored to determine onset, magnitude, and duration of THC intoxication and withdrawal and to correlate with THC and rimonabant pharmacokinetics. Changes in blood oxygen level-dependent (BOLD) signal are determined with five fMRI scans throughout the study. Eighteen non-drug-using controls undergo scanning and cognitive testing at similar intervals.

Risks and Benefits: The proposed doses of THC and rimonabant have been well tolerated in other studies. The most common side effects of oral THC are sedation, cognitive impairment, euphoria, poor coordination, tachycardia, and hypotension. Spontaneous withdrawal from cannabis is mild and medically benign. Experience with other drugs suggests that antagonist-elicited cannabis withdrawal may have an earlier onset and greater intensity than spontaneous cannabis withdrawal. There are no clinical benefits to participants. Scientific benefits are greater understanding of cannabis intoxication, tolerance, and withdrawal and of the role of rimonabant in eliciting cannabis withdrawal.

ELIGIBILITY:
* Eligibility Crtieria for Canabis Users

INCLUSION CRITERIA:

1. 18 to 45 years of age;
2. Cannabis use of at least one year with a typical pattern of daily use for the three months prior to unit admission;
3. A urine sample positive for cannabinoids in the 30 days prior to study enrollment;
4. Blood pressure (BP) and heart rate (HR) at or below the following values while sitting after 5 minutes' rest: Systolic BP (SBP) 140 mm Hg, diastolic BP (DBP) 90 mm Hg,

   heart rate (HR) 100 bpm;
5. 12-lead standard ECG and 3-minute rhythm strip without clinically relevant abnormalities and within the limits defined for the protocol in Appendix 2;
6. Peripheral veins suitable for repeated venipuncture and placement and maintenance of an IV catheter;
7. Ability to swallow capsules;
8. Ability to communicate well with the investigators and to comply with study requirements;
9. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (beta-HCG) pregnancy test prior to study enrollment. All volunteers must use an intra-uterine device or hormonal contraception during the entire study period and for 1 month after. Women who are postmenopausal for more than 12 months or who were sterilized more than 3 months ago are not considered to have childbearing potential;
10. Estimated IQ greater than or equal to 85 determined by the Wechsler Abbreviated Scale of Intelligence
11. Right-handed (Experiment II only).

EXCLUSION CRITERIA:

1. History or presence of any clinically significant disease state, as detected by history, physical examination, and/or laboratory tests, that might put the subject at increased risk of adverse events or that might interfere with the absorption, distribution, metabolism, or excretion of study drugs;
2. Current physical dependence on any substance other than cannabis, nicotine, or caffeine;
3. Positive serological tests for syphilis or HIV infection;
4. Positive purified protein derivative (PPD) test in the absence of a negative chest Xray;
5. Consumption of an investigational drug within 90 days prior to study drug administration;
6. Consumption of any drug at a dose known to have a well-defined potential for toxicity to a major organ system within 3 months prior to study drug administration;
7. Symptoms of a clinically significant1 illness within two weeks prior to study drug administration;
8. History of a clinically significant1 adverse event associated with cannabis intoxication or withdrawal;
9. History of epileptic seizures or head trauma with loss of consciousness greater than three minutes;
10. History of psychosis or any current DSM-IV axis I disorder (other than cannabis, caffeine or nicotine dependence, or simple phobia);
11. Donation of more than 500 mL of blood within 30 days of study drug administration;
12. Regular use of alcohol (greater than or equal to 6 standard drinks per day) four or more times per week in the month prior to study entry;
13. If female, pregnant or nursing;
14. ADHD Screening Rating Scale score greater than or equal to 24 on either the A or B subscale;
15. Allergy to sesame seed oil (ingredient in dronabinol capsules);
16. Currently interested in or participating in drug abuse treatment, or participated in drug abuse treatment within 60 days preceding study enrollment.
17. Claustrophobia that precludes being able to tolerate an fMRI session (Experiment II only).
18. Magnetizable metal on or within the body that cannot be removed (Experiment II only).

Eligibility Criteria for Controls

The goal of the eligibility criteria for control subjects is to obtain a group approximately comparable to the cannabis users in terms of age, sex, ethnicity, and intelligence.

INCLUSION CRITERIA:

1. 18 to 45 years of age;
2. BP and HR at or below the following values while sitting after five minutes' rest: SBP 140 mm Hg, DBP 90 mm Hg, HR 100 bpm;
3. Ability to communicate well with the investigator and to comply with study requirements;
4. If female with reproductive potential, must be using a reliable method of birth control
5. Estimated IQ greater than or equal to 85 determined by the Wechsler Abbreviated Scale of Intelligence;
6. Right-handed

EXCLUSION CRITERIA:

1. History or presence of any clinically significant disease state, as detected by history, physical examination, and/or laboratory tests that might put the subject at increased risk of adverse events;
2. A positive urine test for any illicit drug at any time during screening or study participation;
3. Current physical dependence on any substance other than nicotine or caffeine;
4. Self-reported lifetime use of any illicit drug other than cannabis;
5. Self-reported lifetime use of cannabis greater than ten times or use within the last two years;
6. Positive serological tests for syphilis or HIV infection;
7. History of epileptic seizures or head trauma with loss of consciousness greater than three minutes;
8. History of psychosis or any current DSM-IV axis I disorder (other than caffeine or nicotine dependence, or simple phobia);
9. Regular use of alcohol (greater than or equal to 6 standard drinks per day) four or more times per week in the month prior to study entry;
10. If female, pregnant or nursing;
11. ADHD Screening Rating Scale score greater than or equal to 24 on either the A or B subscale;
12. Claustrophobia that precludes being able to tolerate an fMRI session;
13. Magnetizable metal on or within the body that cannot be removed.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-04-16; Primary Completion 2010-01-11 (Actual); Study Completion 2010-01-11 (Actual)

PRIMARY OUTCOMES:
Determination of the lowest dose of Rimonabant that elicits cannabis withdrawal.

SECONDARY OUTCOMES:
Cognitive, subjective effects, and brain activation after acute and chronic THC and spontaneous antagonist elicited cannabis withdrawal. Rimonabant and THC pharmacokinetics in various biological matrices.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland

REFERENCES:
- [Background] Menzaghi F, Rassnick S, Heinrichs S, Baldwin H, Pich EM, Weiss F, Koob GF. The role of corticotropin-releasing factor in the anxiogenic effects of ethanol withdrawal. Ann N Y Acad Sci. 1994 Oct 31;739:176-84. doi: 10.1111/j.1749-6632.1994.tb19819.x. PMID 7832471
- [Background] Ehrman RN, Robbins SJ, Childress AR, Goehl L, Hole AV, O'Brien CP. Laboratory exposure to cocaine cues does not increase cocaine use by outpatient subjects. J Subst Abuse Treat. 1998 Sep-Oct;15(5):431-5. doi: 10.1016/s0740-5472(97)00290-0. PMID 9751000
- [Background] Copersino ML, Boyd SJ, Tashkin DP, Huestis MA, Heishman SJ, Dermand JC, Simmons MS, Gorelick DA. Cannabis withdrawal among non-treatment-seeking adult cannabis users. Am J Addict. 2006 Jan-Feb;15(1):8-14. doi: 10.1080/10550490500418997. PMID 16449088
- [Derived] Gorelick DA, Goodwin RS, Schwilke E, Schwope DM, Darwin WD, Kelly DL, McMahon RP, Liu F, Ortemann-Renon C, Bonnet D, Huestis MA. Antagonist-elicited cannabis withdrawal in humans. J Clin Psychopharmacol. 2011 Oct;31(5):603-12. doi: 10.1097/JCP.0b013e31822befc1. PMID 21869692